CLINICAL TRIAL: NCT03352271
Title: Comparison of Clinical Outcomes Between Thrice-weekly and Individualized Incremental Hemodialysis in Incident Hemodialysis Patients
Brief Title: Individualized Incremental Hemodialysis Study
Acronym: IIHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Kidney and urology Center (Unknown); Mansoura University (Other); Fasila Hemodialysis Center (Unknown)
Responsible Party: Principal Investigator, Mohamed Elrggal, Principle Investigator, Nephrologist, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MER17MD
Record Dates: First submitted 2017-11-16; First posted 2017-11-24 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Hemodialysis Complication; ESRD; Renal Failure
Keywords: Incremental hemodialysis; Precision medicine; Individualized care
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Incremental hemodialysis (Experimental): ESRD patients starting an individualized (twice/week, once/week, once/10 days or less frequent) incremental hemodialysis program.
  Interventions: Procedure: Individualized Incremental hemodialysis
- Thrice weekly dialysis (Active Comparator): ESRD patients initiating a conventional thrice weekly hemodialysis program
  Interventions: Procedure: Conventional thrice weekly hemodialysis

INTERVENTIONS:
Procedure: Individualized Incremental hemodialysis — Individualized Incremental hemodialysis program (twice/week, once/week, once/10days or less frequent) will be provided to incident ESRD patients according to their symptom presentation, clinical examination, investigations and daily urine volume measurement.
  Arms: Individualized Incremental hemodialysis
Procedure: Conventional thrice weekly hemodialysis — Thrice weekly hemodialysis program, the current standard of care for all patients, as a control
  Arms: Thrice weekly dialysis

SUMMARY:
Thrice weekly hemodialysis has been the standard of care all-over the world for end-stage renal disease (ESRD) requiring renal replacement therapy (RRT). Despite being in the era of precision medicine and individualized healthcare, this program doesn't take into account patients with residual kidney function (RKF) who don't require a thrice weekly hemodialysis frequency. Incremental hemodialysis (defined as twice weekly hemodialysis initiation in incident hemodialysis patients with residual kidney function) has been raised as an alternative to the conventional thrice weekly dialysis. Retrospective trials has proved safety of a twice weekly initiation with comparative efficacy to the thrice weekly program. Despite that, there is paucity of prospective observational and rarity of randomized controlled trials comparing both regimens. In this study, the investigators tend to provide a more individualized incremental hemodialysis approach to incident hemodialysis patients with residual urine volume and RKF. The investigators will compare the results to ESRD patients initiating a thrice weekly hemodialysis program.

DETAILED DESCRIPTION:
This project aims to study the feasibility, safety and efficacy of individualized incremental (twice weekly, once weekly, once/10days or less frequent) hemodialysis (IIHD) initiation versus conventional thrice weekly HD for incident end stage renal disease (ESRD) patients with residual urine volume (RUV > 0.5 L/day, as a reference to residual kidney functions) who chose hemodialysis as their method of renal replacement therapy (RRT).

Incremental HD has been an area of research interest in the past few years with many publications discussing its feasibility and safety for incident HD patients. Smooth transition to dialysis in incident ESRD patients through incremental twice (or even once) weekly dialysis initiation has shown benefits in preservation of residual kidney functions (RKF) in comparison to thrice weekly HD. It has also been proposed as a method of reducing healthcare cost while providing quality healthcare to the patients(1). However, most available data are retrospective analysis, few data are present to compare the results to thrice weekly HD in a randomized controlled or even in a prospective manner. Incremental HD has been also practiced in some parts of Egypt in the last 2-3 years. The investigators will compare outcomes of participants starting a less frequent dialysis program to conventional thrice weekly HD in a multi-center study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage 5 chronic kidney disease (CKD) with estimated glomerular filtration rate of less than 10 ml/min/1.73m2 (using CKD-EPI equation for eGFR).
2. Residual urine volume at least 0.5 L/day or more.

Exclusion Criteria:

1. Children < 18 years of age.
2. Patients who were previously on other types of RRT, either on peritoneal dialysis, or on kidney transplant.
3. Recent (within 3 months) acute kidney injury (AKI).
4. Urine output less than 0.5 L/day.
5. Active malignancy at time of inclusion.
6. Active inflammatory disease with immunosuppressive treatment.
7. Decompensated Liver disease, Hepatorenal syndrome.
8. Cardiovascular disease defined as: heart failure type IV of the New York Heart Association (NYHA) or Cardiorenal syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Survival rate after 24 months | 24 months
  To assess and compare Survival rate after 24 months in incident HD patients with individualized incremental HD (IIHD) as an RRT starting regimen, compared to those patients who start RRT with the conventional thrice weekly method.

SECONDARY OUTCOMES:
All-cause hospitalization rate | 24 months
  Rate of hospital admissions and number of days hospitalized for any cause (including cardiovascular events, CVE) during the 24 months.
Preservation of residual kidney function | 24 months
  Preservation of Residual kidney function (time to anuria defined as urine output UOP < 100 ml/day, rate of decline of RKF defined as the slope in decline of daily UOP measured monthly) during the 24 months of follow up.
Development of hypertrophic cardiomyopathy | 24 months
  Using Echocardiography to detect the development of hypertrophic cardiomyopathy
Cost of care | 24 months
  comparing number of hemodialysis sessions in both groups multiplied by the cost of each session.
Estimation of quality of life (QOL) | 24 months
  Comparing Quality of life survey values from Kidney Disease Quality of Life short form, KDQOL-SF v1.3, Arabic version between each group members
Anemia Profile | 24 months
  Mean hemoglobin levels.
Bone-mineral metabolism profile | 24 months
  Mean levels of calcium, phosphorus, parathyroid hormone PTH
Vascular access complications | 24 months
  rate of infection, thrombosis and hematoma formation

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Elrggal, MD, Principal Investigator — Alexandria University; Mohamed A Sobh, MD, Study Chair — Mansoura University; Hussein A Sheashaa, MD, Study Chair — Mansoura University; Ahmed F Elkeraie, MD, Study Chair — Alexandria University
Locations (2):
- Egypt (2):
  - Mansoura University, Mansourah, Alexandria Governorate
  - kidney and Urology Center, Alexandria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elrggal ME, Zyada R. Gradual initiation of dialysis as a means to reduce cost while providing quality health care. Nat Rev Nephrol. 2017 Nov;13(11):720. doi: 10.1038/nrneph.2017.135. Epub 2017 Sep 25. No abstract available. PMID 28944775
- [Background] Rhee CM, Ghahremani-Ghajar M, Obi Y, Kalantar-Zadeh K. Incremental and infrequent hemodialysis: a new paradigm for both dialysis initiation and conservative management. Panminerva Med. 2017 Jun;59(2):188-196. doi: 10.23736/S0031-0808.17.03299-2. Epub 2017 Jan 13. PMID 28090764
- [Background] Obi Y, Streja E, Rhee CM, Ravel V, Amin AN, Cupisti A, Chen J, Mathew AT, Kovesdy CP, Mehrotra R, Kalantar-Zadeh K. Incremental Hemodialysis, Residual Kidney Function, and Mortality Risk in Incident Dialysis Patients: A Cohort Study. Am J Kidney Dis. 2016 Aug;68(2):256-265. doi: 10.1053/j.ajkd.2016.01.008. Epub 2016 Feb 9. PMID 26867814
- [Background] Obi Y, Eriguchi R, Ou SM, Rhee CM, Kalantar-Zadeh K. What Is Known and Unknown About Twice-Weekly Hemodialysis. Blood Purif. 2015;40(4):298-305. doi: 10.1159/000441577. Epub 2015 Nov 17. PMID 26656764
- [Background] Wong J, Vilar E, Davenport A, Farrington K. Incremental haemodialysis. Nephrol Dial Transplant. 2015 Oct;30(10):1639-48. doi: 10.1093/ndt/gfv231. Epub 2015 Jun 1. PMID 26038351
- [Background] Kalantar-Zadeh K, Unruh M, Zager PG, Kovesdy CP, Bargman JM, Chen J, Sankarasubbaiyan S, Shah G, Golper T, Sherman RA, Goldfarb DS. Twice-weekly and incremental hemodialysis treatment for initiation of kidney replacement therapy. Am J Kidney Dis. 2014 Aug;64(2):181-6. doi: 10.1053/j.ajkd.2014.04.019. Epub 2014 May 17. PMID 24840669
- [Background] Vanholder R, Van Biesen W, Lameire N. Is starting hemodialysis on a twice-weekly regimen a valid option? Am J Kidney Dis. 2014 Aug;64(2):165-7. doi: 10.1053/j.ajkd.2014.06.003. No abstract available. PMID 25060001
- [Background] Rhee CM, Unruh M, Chen J, Kovesdy CP, Zager P, Kalantar-Zadeh K. Infrequent dialysis: a new paradigm for hemodialysis initiation. Semin Dial. 2013 Nov-Dec;26(6):720-7. doi: 10.1111/sdi.12133. Epub 2013 Sep 9. PMID 24016197
- [Background] Libetta C, Esposito P, Dal Canton A. Once-weekly hemodialysis: a single-center experience. Am J Kidney Dis. 2015 Feb;65(2):343. doi: 10.1053/j.ajkd.2014.07.034. No abstract available. PMID 25616635
- [Background] Bieber B, Qian J, Anand S, Yan Y, Chen N, Wang M, Wang M, Zuo L, Hou FF, Pisoni RL, Robinson BM, Ramirez SP. Two-times weekly hemodialysis in China: frequency, associated patient and treatment characteristics and Quality of Life in the China Dialysis Outcomes and Practice Patterns study. Nephrol Dial Transplant. 2014 Sep;29(9):1770-7. doi: 10.1093/ndt/gft472. Epub 2013 Dec 8. PMID 24322579
- [Background] Diao Z, Zhang D, Dai W, Ding J, Zhang A, Liu W. Preservation of residual renal function with limited water removal in hemodialysis patients. Ren Fail. 2011;33(9):875-7. doi: 10.3109/0886022X.2011.605535. Epub 2011 Aug 8. PMID 21819316
- [Background] Elamin S, Abu-Aisha H. Reaching target hemoglobin level and having a functioning arteriovenous fistula significantly improve one year survival in twice weekly hemodialysis. Arab J Nephrol Transplant. 2012 May;5(2):81-6. PMID 22612193
- [Background] Fernandez-Lucas M, Teruel-Briones JL, Gomis-Couto A, Villacorta-Perez J, Quereda-Rodriguez-Navarro C. Maintaining residual renal function in patients on haemodialysis: 5-year experience using a progressively increasing dialysis regimen. Nefrologia. 2012;32(6):767-76. doi: 10.3265/Nefrologia.pre2012.Jul.11517. English, Spanish. PMID 23169359
- [Background] Hanson JA, Hulbert-Shearon TE, Ojo AO, Port FK, Wolfe RA, Agodoa LY, Daugirdas JT. Prescription of twice-weekly hemodialysis in the USA. Am J Nephrol. 1999;19(6):625-33. doi: 10.1159/000013533. PMID 10592355
- [Background] Lin X, Yan Y, Ni Z, Gu L, Zhu M, Dai H, Zhang W, Qian J. Clinical outcome of twice-weekly hemodialysis patients in shanghai. Blood Purif. 2012;33(1-3):66-72. doi: 10.1159/000334634. Epub 2011 Dec 29. PMID 22212562
- [Background] Lin YF, Huang JW, Wu MS, Chu TS, Lin SL, Chen YM, Tsai TJ, Wu KD. Comparison of residual renal function in patients undergoing twice-weekly versus three-times-weekly haemodialysis. Nephrology (Carlton). 2009 Feb;14(1):59-64. doi: 10.1111/j.1440-1797.2008.01016.x. Epub 2008 Nov 19. PMID 19019171
- [Background] Toth-Manikowski SM, Shafi T. Hemodialysis Prescription for Incident Patients: Twice Seems Nice, But Is It Incremental? Am J Kidney Dis. 2016 Aug;68(2):180-183. doi: 10.1053/j.ajkd.2016.04.005. No abstract available. PMID 27477358